CLINICAL TRIAL: NCT01302990
Title: Safety, Tolerability and Immunogenicity of a Plant-Made H1 VLP Influenza Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-H1VLP-003
Record Dates: First submitted 2011-02-11; First posted 2011-02-24 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Flu
Keywords: Influenza; Respiratory disease; Prevention
MeSH Terms: conditions — Influenza, Human; Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 5 micrograms H1 VLP (Experimental)
  Interventions: Biological: Dose given at Day 0
- 13 micrograms H1 VLP (Experimental)
  Interventions: Biological: Dose given at Day 0
- 28 micrograms H1 VLP (Experimental)
  Interventions: Biological: Dose given at Day 0
- 45 micrograms Fluzone (Active Comparator)
  Interventions: Biological: Dose given at Day 0
- Placebo (Placebo Comparator)
  Interventions: Biological: Dose given at Day 0

INTERVENTIONS:
Biological: Dose given at Day 0 — Dose given by intramuscular administration (0.5 mL)

SUMMARY:
This is a Phase 1, randomized, double-blind, active- and placebo-controlled, multicenter, dose-ranging study to evaluate the safety, tolerability and Immunogenicity of a single non-adjuvanted dose of the H1 VLP Influenza vaccine in healthy adults 18-49 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults, 18 to 49 years of age;
* Healthy as judged by the Principal Investigator (PI) or designee and determined by medical history, physical examination, vital signs, screening laboratories and medical history conducted no more than 30 days prior to study vaccine administration;
* BMI of ≥ 18 and ≤ 32;
* Comprehension of the study requirements, expressed availability for the required study period and ability to attend scheduled visits;
* Accessible by telephone on a consistent basis;
* In the opinion of the Investigator, competence and willingness to provide written, informed consent for participation after reading the informed consent form. The subject must have adequate opportunity to discuss the study with an Investigator or qualified designee;
* Showing a HI titer < 1/40 for the swine-origin A/California/07/2009 H1N1-like X-179A strain in sera during the screening period;
* If female and of childbearing potential, have a negative serum pregnancy test result prior vaccination. Female who are post menopausal (no spotting at all) for at least 2 years will not require a pregnancy test;
* If female and capable of childbearing, has been consistently using effective birth control for the 28 days prior to vaccination. An example of highly effective birth control is oral contraceptives, hormone implants, abstinence (confirmed by Investigator), or male condom plus spermicide. All female and of childbearing potential, must provide a serum sample for pregnancy screening. Female of child bearing potential (except subjects in a same sex relationship) must agree to continue employing adequate birth control measures for at least 60 days post vaccination and must have no plan to become pregnant for at least 60 days post vaccination;

Exclusion Criteria:

Presence of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. "Uncontrolled" is defined as:

1. Requiring a new medical or surgical treatment within one month prior to study vaccine administration;
2. Requiring a change in medication dosage in one month prior to study vaccine administration due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable), or
3. Hospitalization or an event fulfilling the definition of a serious adverse event within one month prior to study vaccine administration;

   * Any medical or neuropsychiatric condition or any history of excessive alcohol use or drug abuse which, in the Investigator's opinion, would render the subject incompetent to provide informed consent or unable to provide valid safety observations and reporting;
   * Any confirmed or suspected immunosuppressive condition or immunodeficiency including history of human immunodeficiency virus (HIV) infection, Hepatitis B or C, or the presence of lymphoproliferative disease;
   * Presence of any febrile illness, oral temperature of > 38.0˚C (100.4˚F) within 24 hours prior to randomization. Such subjects may be re-evaluated for randomization after resolution of illness;
   * History of autoimmune disease;
   * Administration of any vaccine (including any other influenza vaccine) within a 30 day period prior to study enrollment, or planned administration within the period from the first vaccination up to blood sampling at Day 21 or within 30 days prior to blood sampling at Day 201. Immunization on an emergency basis of a tetanus and diphtheria toxoids adsorbed for adult use (Td) will be allowed provided the vaccine is not administered within two weeks prior to study vaccine administration. Receipt of any other emergency immunizations (e.g. rabies) will result in a case-by-case review by the medical monitor of continued participation;
   * Use of any investigational or non-marketed product within 30 days prior to study enrollment or planned use during the study period. Subjects may not participate in any other investigational or marketed drug study while participating in this study;
   * Treatment with systemic glucocorticoids at a dose exceeding 10 mg of prednisone per day, or equivalent for more than 7 consecutive days or for 10 or more days in total, within one month of first study vaccine administration, or any other cytotoxic or immunosuppressant drug within three months of vaccination.
   * Use of any immune globulin product
   * Use of high dose inhaled steroids or oral and parenteral high dose steroid medications. Nasal steroids are allowed. Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving prophylactic anti-platelet medications, e.g., low-dose aspirin [eg</= 325 mg/day (1 regular adult aspirin) or </= 81 mg/day (1 baby aspirin)], and without a clinically apparent bleeding tendency are eligible;
   * History of allergy to any of the constituents of H1 VLP (H1N1) study vaccine, or the phosphate buffer;
   * History of allergy to egg-based vaccines such as allergy or hypersensitivity to egg proteins.
   * History of severe allergic reactions or anaphylaxis or severe asthma;
   * History of tobacco allergy;
   * History of anti-histaminics used continuously for 4 weeks or more at any time in the past year, prior to randomization;
   * Have a rash, dermatological condition or tattoos which may interfere with injection site reaction rating;
   * Have received a blood transfusion within 90 days prior to vaccination;
   * If female, either known pregnancy or urine beta-human chorionic gonadotropin (ß-hCG) test results consistent with pregnancy during the screening period and prior to study vaccine administration on Day 0;
   * Female subjects who are lactating;
   * Any vital sign abnormalities: systolic blood pressure, diastolic blood pressure, resting pulse rate or not well controlled and according to the Investigator's opinion;
   * Cancer or treatment for cancer within 3 years of study vaccine administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible.
   * Subject with a history of Gillian Barre Syndrome

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Percentage, intensity and relationship of immediate complaints, 30 minutes post-vaccination Percentage, intensity and relationship of immediate complaints, 30 minutes post-vaccination as a measure of safety and tolerability | 30 minutes after vaccination
Percentage, intensity and relationship to vaccination of solicited local and systemic signs and symptoms as a measure of safety and Tolerability | 7 days after vaccination
Percentage, intensity and relationship of solicited and unsolicited local and systemic signs and symptoms 21 days following a single dose of study vaccine as a measure of safety and tolerability | 21 days after vaccination
Occurrences of all adverse events, and serious adverse events during the study as a measure of safety and Tolerability | 6 months
Occurrences of new onset of a chronic disease (NOCD)during the study as a measure of safety and tolerability | 6 months
The number and percentage of subjects with normal and abnormal urine, haematological and biochemical values at Screening, Days 21 and 201 as a measure of safety and tolerability | 6 months

SECONDARY OUTCOMES:
Immunogenicity | 21 days and 6-month after injection
  Specific antibodies: Geometric Mean Titers (GMTs) with 95% confidence interval by using the Hemagglutination-Inhibition (HI), MicroNeutralisation (MN) and the Single Radial Hemolysis (SRH) tests; To measure the increase in antibodies directed to plant-specific glycans.

CONTACTS AND LOCATIONS:
Overall Officials: William E Gannon, MD, Principal Investigator — Accelovance
Locations (1):
- Accelovance, Rockville, Maryland, United States